CLINICAL TRIAL: NCT04084691
Title: Capillary Glycerolemia Evolution During Physical Exercise
Acronym: LSEEGLYCEROL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 190089 - IDRCB 2019-A00200-57
Record Dates: First submitted 2019-08-01; First posted 2019-09-10 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2020-11

CONDITIONS: Physical Activity; Body Mass Index
MeSH Terms: conditions — Motor Activity | interventions — Angptl4 protein, mouse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Every patient will undergo every combination of physical exercise/meal type (3x3 combinations), one following the other. Each combination is replicated three times.
  Interventions: Other: Physical exercice - moderate intensity; Other: Physical exercice - high intensity; Other: Physical exercice - workout; Other: Normal meal; Other: Normalized meal; Other: Fasting

INTERVENTIONS:
Other: Physical exercice - moderate intensity — standardized physical activity (moderate intensity) lasting 30 minutes and having a warm-up portion of 5 minutes
Other: Physical exercice - high intensity — standardized physical activity (high intensity) lasting 30 minutes and having a warm-up portion of 5 minutes
Other: Physical exercice - workout — standardized physical activity (bodybuilding) lasting 30 minutes and having a warm-up portion of 5 minutes
Other: Normal meal — - Hyperlipidic meal Energy supply: 800 kcal Distribution of macronutrients: proteins: 15% +/- 5; carbohydrates: 40% +/- 5; lipids: 45 +/- 5 Choice of foods determined with the dietician taking into account the patient's tastes and products available on the market The same meal will be taken before the 3 sessions concerned.
Other: Normalized meal — - Hyperglucidic meal Energy supply: 800 kcal Macronutrient distribution: protein 15% +/- 5; carbohydrates 60% +/- 5; lipids 25 +/- 2 Choice of foods determined with the dietician taking into account the patient's tastes and products available on the market.
  The same meal will be taken before the 3 sessions concerned.
Other: Fasting — non meal in the hour before exercise

SUMMARY:
Maximum fatty acid oxidation is known to occur at exercise intensities between 45 and 65% VO2max and in the fasting state.

However, the optimal level may depend on various unknown factors. Glycerolemia is a good marker of the fatty acid metabolism but its evolution remains poorly described, maybe due to the difficulty of the measure.

A new device allows an easy measurement of glycerolemia during exercise and could enable personalization strategies to optimize exercise efficacy.

In this study, the investigators plan to test three different exercise types and three different fasting conditions with three replicates each to evaluate the variability of glycerolemia and its evolution during exercise.

DETAILED DESCRIPTION:
The metabolism of mobilized fatty acids as an energy reserve during physical exercise produces glycerol, which makes it a marker of the intensity of lipolysis.

This measurement of the intensity of lipolysis in humans can be carried out according to several methods. Since glycerol is a product of lipolysis, its rate of appearance (Ra) in the blood represents a physical quantity naturally associated with lipolysis activity. Unfortunately, its quantification requires the use of a tracer isotope (deuterated glycerol), which limits its applicability. The alternative is the determination of glycerolemia in the blood or in the interstitial fluid via a microdialysis probe placed in subcutaneous adipose tissue;

Recently, a measuring device has been proposed which makes it possible to measure glycerolemia from capillary blood, in the manner of measuring blood glucose in diabetic patients. This device has the advantage of being used repeatedly after a physical exercise. This flexibility also makes it possible to consider the personalization of the sports program by identifying the circumstances associated with an increase in lipolysis such as the type of meal preceding the exercise or its intensity.

Evidence suggests that moderate-intensity exercise (about 45% -65% VO2max) performed under fasting conditions maximizes lipid metabolism as a source of energy, compared with carbohydrate metabolism. But these data conceal a likely significant variability in individual outcomes, including levels of training, gender, age, and nutritional intake prior to exercise. Our hypothesis is that the current recommendation to the diabetic patient, or with a metabolic syndrome, to exercise moderate intensity fasting physical activity could be adapted individually to each patient in order to optimize the benefits of such a practice. In this sense, the easy access to a measurement of capillary glycerolemia could make it possible to identify in a personalized way the type of physical activity.

This research project aims to accurately describe the evolution of capillary glycerolemia in several configurations of physical exercise (variable intensity) by controlling the effect of the previous meal. It will also seek to identify situations associated with a greater increase in capillary glycerolemia to pave the way for personalization of the sports activity program.

ELIGIBILITY:
Inclusion criteria :

* Major patients followed in Diabetology-Nutrition Day Hospital of Bichat-Claude Bernard Hospital as part of the ETAPES program
* overweight or obese patient: body mass index BMI> 25 kg / m²
* Volunteer to participate in and follow a proposed physical activity program as part of regular follow-up
* Volunteer to participate in the research, comfortable with the use of the device of auto measurement of capillary glycerolemia

Exclusion criteria :

* Pregnancy in progress or breastfeeding
* Patient under guardianship or curatorship
* Patient participating in another interventional research protocol
* No affiliation to the social security scheme or French Universal Health Cover (CMU)
* Absence of informed consent, written and signed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-10-23 (Actual); Primary Completion 2020-09-11 (Actual); Study Completion 2020-09-11 (Actual)

PRIMARY OUTCOMES:
concentration of glycerol in capillary blood | at the beginning of exercise
  The primary endpoint is the time series of measurements of capillary glycerol concentration using the DietSee device (LSEE, Ajaccio, France)
concentration of glycerol in capillary blood | 20 minutes after the beginning of exercise
  The primary endpoint is the time series of measurements of capillary glycerol concentration using the DietSee device (LSEE, Ajaccio, France)
concentration of glycerol in capillary blood | 30 minutes after the beginning of exercise
  The primary endpoint is the time series of measurements of capillary glycerol concentration using the DietSee device (LSEE, Ajaccio, France)
concentration of glycerol in capillary blood | 45 minutes after the beginning of exercise
  The primary endpoint is the time series of measurements of capillary glycerol concentration using the DietSee device (LSEE, Ajaccio, France)
concentration of glycerol in capillary blood | 60 minutes after the beginning of exercise
  The primary endpoint is the time series of measurements of capillary glycerol concentration using the DietSee device (LSEE, Ajaccio, France)

SECONDARY OUTCOMES:
1. Maximum concentration of glycerol in capillary blood | from the beginning of the exercise and during one hour
  Maximum capillary glycerolemia (peak) among the time series
2. Glycerol concentration in peripheral venous blood, | 30 minutes after the beginning of bodybuilding exercise (i.e. at the end of the exercice)
  Glycerolemia in peripheral venous blood, measured at the end of a bodybuilding type exercise session

CONTACTS AND LOCATIONS:
Overall Officials: Boris HANSEL, MD PHD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Bichat Claude-Bernard, Paris, France

IPD SHARING:
Plan to Share IPD: No